CLINICAL TRIAL: NCT01869855
Title: Use of Subperiosteal Drainage Versus Subdural Drainage in Chronic Subdural Hematomas Treated With Burr-Hole Trepanation: a Randomized Controlled Trial
Brief Title: A Prospective Randomized Study Evaluating the Recurrence Rate of Chronic Subdural Hematoma After Placing a Subperiosteal Drainage Compared to a Subdural Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Dr. Jehuda Soleman, MD, Kantonsspital Aarau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSDH-KSA
Record Dates: First submitted 2013-06-02; First posted 2013-06-05 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Chronic Subdural Hematoma
Keywords: chronic subdural hematoma; traumatic brain injury; burr hole trepanation; drainage after evacuation of chronic subdural hematoma; intracranial bleed
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Brain Injuries, Traumatic; Intracranial Hemorrhages

ARMS (2):
- 110 patients with cSDH assigned to subdural drainage (Active Comparator): Randomization of 110 patients with cSDH to one treatment group (subdural or subperiosteal drainage) out of the 220 patients included in the study.
  Interventions: Procedure: Subdural Drainage
- 110 patients with cSDH assigned to subperiosteal drainage (Active Comparator): Randomization of 110 patients with cSDH to one treatment group (subdural or subperiosteal drainage) out of the 220 patients included in the study.
  Interventions: Procedure: Subperiosteal Drainage

INTERVENTIONS:
Procedure: Subdural Drainage
  Arms: 110 patients with cSDH assigned to subdural drainage
Procedure: Subperiosteal Drainage
  Arms: 110 patients with cSDH assigned to subperiosteal drainage

SUMMARY:
The aim of our study is to investigate in randomized controlled fashion whether the recurrence and complication rate, after insertion of subperiosteal drainage in the treatment of chronic subdural haematoma, is higher compared to insertion of subdural drainage.

We hypothesize that patients treated with a subperiosteal drainage do not show higher recurrence rates than those treated with a subdural drainage, and suffer less complications.

DETAILED DESCRIPTION:
Chronic subdural haematoma (cSDH) is one of the most frequent neurosurgical entities, affecting elderly people and associated with substantial morbidity and mortality. Its incidence is reported to be 1.7-13.1 per 100000 inhabitants per year, yet there has been a steady increasing incidence as the result of prolonged life expectancy in recent years. Surgical treatment is recommended in case of neurological symptoms. In the only evidence based review of the different surgical treatment modalities of cSDH, Weigels study group concluded that bure-hole craniostomy with irrigation and drainage has the best cure to complication ratio. A randomized controlled study of Santarius and his colleagues showed a reduced recurrence and mortality while placing a subdural drainage compared to no drainage after burr hole evacuation of cSDH. Gazzeri et al. and Zumofen et al. used closed subperiosteal drainage instead of the commonly used subdural drainage. They showed equal or superior results in outcome, complications and postoperative symptoms compared to previous studies. Since the subperiosteal drainage is not positioned in direct contact to cortical structures, bridging veins or haematoma membranes it is considered safer and should be favored over a subdural drainage. Bellut et al. compared in their institute retrospectively 48 patients treated with subperiosteal drainage to 65 patients with subdural drainage and found no difference in recurrence rate of cSDH, yet less mortality and fewer serious complications in the group treated with subperiosteal drainage. However in their study none of the results showed a significant difference, and they concluded that further randomized studies with larger patient number are needed. In a recently published prospective randomized study Kaliaperumal et al. concluded that the recurrence rate in subperiosteal drainage is equal to subdural drainage, yet the modified ranking scale(mRS) of the patients with subperiosteal drainage after 6 months was significantly better. However, the mRS score preoperative were better in the subperiosteal drain group causing a statistical bias. In addition the amount patients studied was small (25 per group) and the recurrence rate was overall at 0%, with a very low morbidity and mortality compared to the literature. Due to these bias the authors recommend further prospective and randomized studies with larger group of patients.

To date in neurosurgery practice evidence based guidelines on which drainage should be used in cSDH do not exist and both methods, subdural drainage and subperiosteal drainage, are being practiced, depending on the institute and/or the practicing neurosurgeon.

The aim of our study is to investigate in randomized controlled fashion whether the recurrence and complication rate, after insertion of subperiosteal drainage in the treatment of chronic subdural haematoma, is higher compared to insertion of subdural drainage.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age presenting with a symptomatic chronic subdural hematoma
* Chronic subdural hematoma verified on cranial CT or MRI

Exclusion Criteria:

* The surgeon decides based on intraoperative conditions to perform a craniotomy (e.g. acute hematoma indicating a craniotomy)
* Chronic subdural hematoma caused by another underlying illness (e.g. caused by over-drainage of a vp-shunt)
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Recurrence Rate | within the first 12 months postoiperatively

SECONDARY OUTCOMES:
Complication rate (Morbidity) | within the first 12 months postoperatively
Mortality | within the first 12 months postoperatively
Outcome: Markwalder Score | within the first 12 months postoperatively
Outcome: modified Ranking Score | within the first 12 months postoperatively
Outcome: Glasgow Outcome Score | within the first 12 months postoperatively

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Neurosurgery Kantonsspital Aarau, Aarau, Canton of Aargau
  - Neurosurgery University Hospital of Basel, Basel

REFERENCES:
- [Derived] Soleman J, Lutz K, Schaedelin S, Mariani L, Fandino J. Use of Subperiosteal Drain Versus Subdural Drain in Chronic Subdural Hematomas Treated With Burr-Hole Trepanation: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2016 Apr 8;5(2):e38. doi: 10.2196/resprot.5339. PMID 27059872